CLINICAL TRIAL: NCT04630158
Title: A 12-week Parallel Group, Randomized, Placebo-controlled, Double-blinded, Multi-center Study to Evaluate Efficacy and Safety of 2 Concentrations of SAF312 Eye Drops (5 mg/ml and 15 mg/ml) Used Twice-daily in the Treatment of Post-operative Corneal Induced Chronic Pain (CICP) Following Photorefractive Keratectomy (PRK) or Laser-assisted in Situ Keratomileusis (LASIK) Surgeries
Brief Title: Study of Efficacy and Safety of SAF312 Eye Drops in Subjects With Post-operative Corneal Induced Chronic Pain (CICP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSAF312B12201; 2021-005857-97 (EudraCT Number)
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Chronic Ocular Pain
Keywords: Eye pain; Dry eye like symptoms; Ocular surface pain; Corneal induced chronic pain; neuropathic eye pain; post-operative corneal induced chronic pain; CICP; corneal; corneal pain
MeSH Terms: conditions — Eye Pain | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAF312 Placebo (Placebo Comparator): Randomized to a 1:1:1 topical eye drops, twice daily
  Interventions: Other: SAF312 Placebo
- SAF312 5 mg/mL (Experimental): Randomized to a 1:1:1 topical eye drops, twice daily
  Interventions: Drug: SAF312
- SAF312 15 mg/mL (Experimental): Randomized to a 1:1:1 topical eye drops, twice daily
  Interventions: Drug: SAF312

INTERVENTIONS:
Other: SAF312 Placebo — Topical ocular, suspension eye drops
  Other Names: Artificial tears
  Arms: SAF312 Placebo
Drug: SAF312 — Topical ocular, suspension eye drops
  Arms: SAF312 15 mg/mL; SAF312 5 mg/mL

SUMMARY:
The study was designed to demonstrate the safety and efficacy of two dose concentrations of SAF312 eye drops (5 mg/mL and 15 mg/mL) in subjects with CICP persisting at least for 4 months after refractive or cataract surgery and chronicity confirmed during the observational period. The study also determined the optimal dose to carry forward for further development.

DETAILED DESCRIPTION:
This was a Phase II randomized, double-masked, multi-center, parallel group, placebo-controlled study to evaluate the safety and efficacy of SAF312, 5 mg/mL and 15 mg/mL eye drops versus Placebo used twice-daily in both eyes for 12 weeks. The study consisted of a 12-week observation period starting from Screening Visit (Visit 1) until the Baseline/Randomization Visit (Visit 2). Subjects who met eligibility criteria at Visit 2 were randomized to one of the three treatment arms (SAF312 5 mg/mL, SAF312 15 mg/mL, Placebo) in a 1:1:1 ratio. Subjects who qualified for randomization had visits every 2 weeks for the first 4 weeks, and then monthly visits for the remainder of the 12-week treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who have undergone refractive surgery (i.e., PRK, LASIK, LASEK, RK, or SMILE) in both eyes or cataract surgery in both eyes, with or without refractive enhancement in one or both eyes, ≥4 months prior to Screening Visit and experiencing persistent ocular surface pain since the surgery, and have been seen by an ophthalmologist or optometrist at least once with complaint of continued ocular pain since surgery.
* Subjects who demonstrate a ≥ 60% reduction in ocular pain within 5 minutes after instillation of a single topical ocular anesthetic drop at Screening Visit.

At Baseline

* Subjects with an average pain severity VAS score of ≥ 30 mm based on Daily eDiary for the last 7 days prior to Baseline Visit.
* Subjects who have reported pain severity >10 mm based on Daily eDiary for > 50% of the days of the observational period (Screening)

Key Exclusion Criteria:

* Use of nerve growth factor eye drops within 14 days of the Screening Visit
* Seasonal allergic conjunctivitis, or other acute or seasonal ocular diagnosis that are active at the time of Screening or would be active during the course of the study.
* Any history of ocular herpes simplex virus or herpes zoster virus infection, or other severe ocular conditions such as graft versus host disease, Stevens-Johnson syndrome or sarcoidosis.
* Presence of any ocular infection (bacterial, viral, or fungal) within 30 days prior to Screening.
* Chronic topical ocular medications (ie. cyclosporine, lifitegrast) initiated <6 months prior to Screening Visit, or any anticipated change during the study.
* Use of ocular or nasal corticosteroids within 30 days of Screening Visit.
* Use of neuromodulatory medications (eg, gabapentin, pregabalin) or opioid use for non-ocular pain within 30 days of Screening Visit.
* Chronic medications (both over the counter and prescription) that have not been stable for at least 30 days prior to Screening Visit, or any anticipated change in the chronic medication regimen.
* Subjects requiring hospitalization within 6 months prior to screening for severe psychiatric disorders (e.g. psychosis, schizophrenia, mania, depression) or major psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (22):
  - North Valley Eye Medical Group, Mission Hills, California
  - NVISION Eye Centers, Newport Beach, California
  - Stanford Eye Laser Center, Palo Alto, California
  - Gordon Schanzlin New Vision Inst, San Diego, California
  - Novartis Investigative Site, Coral Springs, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Sight, Needham, Massachusetts
  - Univ of MI Kellogg Eye Center ., Ann Arbor, Michigan
  - Duke Univ Medical Center Ophthalmology, Durham, North Carolina
  - Bergstrom Eye Research LLC, Fargo, North Dakota
  - University of Pennsylvania ., Philadelphia, Pennsylvania
  - Chattanooga Eye Institute, Chattanooga, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Advancing Vision Research LLC, Smyrna, Tennessee
  - Novartis Investigative Site, Houston, Texas
  - Lake Travis Eye and Laser Ctr, Lakeway, Texas
  - Stacy R Smith MD PC, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Rainier Clinical Research Center Inc ., Renton, Washington
  - Periman Eye Institute, Seattle, Washington
- Japan (2):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Shinagawa, Tokyo
- United Kingdom (2):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAF312 15 mg/mL | SAF312 5 mg/mL | SAF312 Placebo
Started | 50 | 49 | 51
Completed | 46 | 45 | 47
Not Completed | 4 | 4 | 4
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAF312 15 mg/mL | SAF312 5 mg/mL | SAF312 Placebo | Total
Number analyzed (Participants) | 50 | 49 | 51 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (15.56) | 60.4 (15.12) | 56.8 (17.15) | 59.4 (15.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 40 | 109
  Male | 15 | 15 | 11 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6
  Not Hispanic or Latino | 47 | 49 | 48 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 7 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 6 | 5 | 4 | 15
  White | 35 | 37 | 38 | 110
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 in Ocular Pain Severity Visual Analog Scale (VAS)
Description: The pain severity Visual Analogue Scale (VAS) was completed by the subject using an electronic diary. A vertical mark was placed on the horizontal scoring line (anchored with 'No Pain' on the left and 'Very Severe' pain on the right) to score the severity of ocular pain over the past 24 hours, with a range from 0 (min) to 100 (max). Higher scores indicate higher pain severity. A negative change from baseline is a positive outcome.
Time Frame: Baseline, Week 12
Population: Full Analysis Set - all treated patients
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- SAF312 5mg/mL; SAF312 Placebo: Randomized to a 1:1:1 topical eye drops, twice daily
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 50 | 49 | 51
Scores on a scale | -23.7 (3.70) | -21.7 (3.71) | -25.3 (3.51)
Statistical Analysis 1: Comparison: SAF312 15 mg/mL vs SAF312 Placebo; Test type: Superiority; p = 0.930, Mixed Models Analysis — Reporting the adjusted p-value derived based on Dunett procedure; mixed-model repeated measures (MMRM) analysis; Least Square (LS) mean difference = 1.6, 95% CI 2-sided [-8.5 to 11.7], Standard Error of Mean 5.10
Statistical Analysis 2: Comparison: SAF312 5mg/mL vs SAF312 Placebo; Test type: Superiority; p = 0.699, Mixed Models Analysis — Reporting the adjusted p-value derived based on Dunett procedure; mixed-model repeated measures (MMRM) analysis; Least Square (LS) mean difference = 3.7, 95% CI 2-sided [-6.4 to 13.8], Standard Error of Mean 5.11

2. Secondary Outcome: Ocular Pain Severity Visual Analog Scale (VAS): Summary Statistics of Change From Baseline at Day 7 and Day 14
Description: as for outcome 1
Time Frame: Baseline, Days 7 and 14
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 45 | 44 | 44
Scores on a scale
  Day 7 (n=45,44,43): number analyzed (Participants) | 45 | 44 | 43
  Day 7 (n=45,44,43) | -10.89 (18.373) | -11.45 (20.661) | -17.40 (21.558)
  Day 14 (n=45,37,44): number analyzed (Participants) | 45 | 37 | 44
  Day 14 (n=45,37,44) | -12.20 (21.484) | -14.89 (25.790) | -21.00 (21.624)

3. Secondary Outcome: Ocular Pain Frequency Visual Analog Scale (VAS): Summary Statistics of Weekly Mean Change From Baseline to Week 12
Description: The pain frequency Visual Analogue Scale (VAS) was completed by the subject using an electronic diary. A vertical mark was placed on the horizontal scoring line (anchored with 'No Pain' on the left and 'Very Frequent' pain on the right) to score the frequency of ocular pain over the past 24 hours, with a range from 0 (min) to 100 (max). Higher scores indicate higher pain frequency. A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 1 to 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 50 | 49 | 50
Scores on a scale
  Week 1 | -10.22 (16.404) | -9.96 (15.464) | -12.45 (15.484)
  Week 2 (n=49,48,50): number analyzed (Participants) | 49 | 48 | 50
  Week 2 (n=49,48,50) | -14.38 (21.073) | -12.68 (20.344) | -18.80 (20.489)
  Week 3 (n=49,47,49): number analyzed (Participants) | 49 | 47 | 49
  Week 3 (n=49,47,49) | -17.35 (21.332) | -14.75 (23.314) | -22.45 (22.980)
  Week 4 (n=49,46,48): number analyzed (Participants) | 49 | 46 | 48
  Week 4 (n=49,46,48) | -19.06 (23.070) | -12.75 (24.076) | -24.07 (25.230)
  Week 5 (n=49,46,48): number analyzed (Participants) | 49 | 46 | 48
  Week 5 (n=49,46,48) | -20.34 (24.524) | -14.31 (23.711) | -26.18 (22.404)
  Week 6 (n=48,47,48): number analyzed (Participants) | 48 | 47 | 48
  Week 6 (n=48,47,48) | -19.84 (25.511) | -15.60 (23.332) | -23.88 (25.433)
  Week 7 (n=47,47,48): number analyzed (Participants) | 47 | 47 | 48
  Week 7 (n=47,47,48) | -22.84 (25.774) | -17.60 (24.715) | -25.09 (24.489)
  Week 8 (n-47,45,48): number analyzed (Participants) | 47 | 45 | 48
  Week 8 (n-47,45,48) | -23.25 (26.009) | -17.40 (23.636) | -24.69 (26.072)
  Week 9 (n=46,44,48): number analyzed (Participants) | 46 | 44 | 48
  Week 9 (n=46,44,48) | -24.30 (25.650) | -18.01 (25.040) | -24.92 (25.648)
  Week 10 (n=46,44,47): number analyzed (Participants) | 46 | 44 | 47
  Week 10 (n=46,44,47) | -25.16 (25.381) | -18.44 (24.387) | -25.72 (26.428)
  Week 11 (n=46,45,47): number analyzed (Participants) | 46 | 45 | 47
  Week 11 (n=46,45,47) | -26.62 (26.057) | -21.68 (24.754) | -25.66 (28.343)
  Week 12 (n=46,43,47): number analyzed (Participants) | 46 | 43 | 47
  Week 12 (n=46,43,47) | -26.24 (25.322) | -20.38 (24.296) | -26.98 (25.977)

4. Secondary Outcome: Ocular Pain Assessment Scale (OPAS) Subscale Quality of Life: Summary Statistics of Change From Baseline to Week 12
Description: Each question in the Ocular Pain Assessment Survey (OPAS) quality of life subscale was scored by the subject on a line marked from 0 (not at all) to 10 (completely) that described how much pain interfered with or affected a particular activity (max score= 10/question). A higher score suggests a higher impact by pain on a particular activity. A negative change from baseline is a positive outcome. There are 7 questions in total regarding Quality of Life. The average score of the 7 Quality of Life questions is reported (mean (SD)).
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 48 | 46 | 49
Scores on a scale
  Week 2 (n=48,46,46): number analyzed (Participants) | 48 | 46 | 46
  Week 2 (n=48,46,46) | -1.39 (1.839) | -0.99 (2.027) | -1.52 (1.704)
  Week 4 (n=46,46,49): number analyzed (Participants) | 46 | 46 | 49
  Week 4 (n=46,46,49) | -1.68 (2.360) | -1.39 (2.040) | -2.00 (2.138)
  Week 8 (n=47,45,45): number analyzed (Participants) | 47 | 45 | 45
  Week 8 (n=47,45,45) | -1.61 (2.428) | -1.30 (2.103) | -1.82 (1.805)
  Week 12 (n=45,45,45): number analyzed (Participants) | 45 | 45 | 45
  Week 12 (n=45,45,45) | -2.20 (2.317) | -1.79 (2.225) | -2.06 (2.284)

5. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Redness - Nasal (Oculus Dexter (OD) = Right Eye)
Description: Conjunctival redness in each of two regions (nasal and temporal) was graded on a scale from 0 to 5 using the McMonnies conjunctival redness photographic scale (max score=5/region). Higher scores suggest higher degrees of redness (worsening). A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | -0.1 (0.75) | -0.0 (0.43) | -0.1 (0.65)
  Week 4 (n=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (n=44,45,46) | -0.2 (0.77) | -0.0 (0.67) | 0.0 (0.52)
  Week 8 (n=45,43,42): number analyzed (Participants) | 45 | 43 | 42
  Week 8 (n=45,43,42) | -0.2 (0.72) | -0.1 (0.68) | -0.2 (0.62)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | -0.2 (0.70) | -0.0 (0.75) | -0.1 (0.76)

6. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Redness - Nasal (Oculus Sinister (OS) = Left Eye)
Description: as for outcome 5
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | -0.2 (0.67) | -0.1 (0.45) | -0.2 (0.61)
  Week 4 (N=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (N=44,45,46) | -0.3 (0.78) | 0.0 (0.67) | -0.1 (0.41)
  Week 8 (n=45,43,42): number analyzed (Participants) | 45 | 43 | 42
  Week 8 (n=45,43,42) | -0.2 (0.70) | -0.2 (0.73) | -0.2 (0.61)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | -0.2 (0.68) | -0.1 (0.59) | -0.2 (0.83)

7. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Redness - Temporal (Oculus Dexter (OD) = Right Eye)
Description: The pain severity Visual Analogue Scale (VAS) was completed by the subject using an electronic diary. A vertical mark was placed on the horizontal scoring line (anchored with 'No Pain' on the left and 'Very Severe' pain on the right) to score the severity of ocular pain over the past 24 hours, with a range from 0 (min) to 100 (max). Higher scores indicate higher pain severity. A negative change from baseline is a positive outcome. A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | -0.2 (0.72) | 0.1 (0.55) | -0.1 (0.68)
  Week 4 (n=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (n=44,45,46) | -0.3 (0.83) | 0.0 (0.71) | -0.1 (0.57)
  Week 8 (n=45,43,42): number analyzed (Participants) | 45 | 43 | 42
  Week 8 (n=45,43,42) | -0.2 (0.84) | -0.1 (0.80) | -0.2 (0.76)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | -0.3 (0.78) | -0.1 (0.73) | -0.3 (0.99)

8. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Redness - Temporal (Oculus Sinister (OS) = Left Eye)
Description: as for outcome 5
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | -0.2 (0.74) | 0.0 (0.53) | -0.1 (0.72)
  Week 4 (n=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (n=44,45,46) | -0.4 (0.81) | 0.1 (0.61) | 0.1 (0.57)
  Week 8 (n=45,43,42): number analyzed (Participants) | 45 | 43 | 42
  Week 8 (n=45,43,42) | -0.2 (0.67) | -0.1 (0.70) | -0.1 (0.69)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | -0.3 (0.71) | -0.1 (0.63) | -0.2 (0.90)

9. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Staining (Oculus Dexter (OD) = Right Eye)
Description: The degree of lissamine conjunctival staining in two regions (temporal and nasal) was graded on a scale from 0 to 4 (max score = 8/eye). Higher scores suggest higher degrees of corneal staining (worsening). A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | 0.1 (0.99) | -0.0 (1.23) | -0.1 (1.06)
  Week 4 (n=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (n=44,45,46) | 0.0 (1.27) | 0.2 (1.62) | -0.2 (1.23)
  Week 8 (n=45,42,42): number analyzed (Participants) | 45 | 42 | 42
  Week 8 (n=45,42,42) | -0.2 (1.00) | 0.0 (1.06) | 0.3 (1.27)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | 0.1 (1.39) | -0.1 (1.24) | 0.0 (1.54)

10. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Conjunctival Staining (Oculus Sinister (OS) = Left Eye)
Description: as for outcome 9
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 47 | 45 | 46
Scores on a scale
  Week 2 (n=47,44,43): number analyzed (Participants) | 47 | 44 | 43
  Week 2 (n=47,44,43) | 0.0 (0.99) | -0.1 (1.51) | -0.2 (1.41)
  Week 4 (n=44,45,46): number analyzed (Participants) | 44 | 45 | 46
  Week 4 (n=44,45,46) | -0.1 (1.20) | 0.1 (1.47) | -0.1 (1.41)
  Week 8 (n=45,42,42): number analyzed (Participants) | 45 | 42 | 42
  Week 8 (n=45,42,42) | -0.2 (1.01) | -0.3 (1.32) | 0.1 (1.46)
  Week 12 (n=44,43,44): number analyzed (Participants) | 44 | 43 | 44
  Week 12 (n=44,43,44) | -0.1 (1.25) | -0.1 (1.16) | -0.1 (1.25)

11. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Corneal Staining (Oculus Dexter (OD) = Right Eye)
Description: The degree of corneal fluorescein staining in each of five regions (superior, inferior, nasal, temporal, and central) was graded on a scale from 0 to 4 (max score=20/eye). Higher scores suggest higher degrees of corneal staining (worsening). A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 49 | 47 | 49
Scores on a scale
  Week 2 (n=49,46,46): number analyzed (Participants) | 49 | 46 | 46
  Week 2 (n=49,46,46) | -0.6 (2.02) | -0.7 (1.73) | -0.7 (2.76)
  Week 4 (n=46,47,49): number analyzed (Participants) | 46 | 47 | 49
  Week 4 (n=46,47,49) | -0.8 (2.84) | -0.1 (2.47) | -0.9 (2.32)
  Week 8 (n=47,45,45): number analyzed (Participants) | 47 | 45 | 45
  Week 8 (n=47,45,45) | -0.9 (2.93) | -0.6 (2.09) | -0.8 (2.40)
  Week 12 (n=46,45,47): number analyzed (Participants) | 46 | 45 | 47
  Week 12 (n=46,45,47) | -0.7 (3.10) | -0.1 (1.95) | -1.5 (2.78)

12. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week - Corneal Staining (Oculus Sinister (OS) = Left Eye)
Description: as for outcome 11
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 49 | 47 | 49
Scores on a scale
  Week 2 (n=49,46,46): number analyzed (Participants) | 49 | 46 | 46
  Week 2 (n=49,46,46) | -0.5 (2.48) | -0.7 (2.55) | -1.0 (2.82)
  Week 4 (n=46,47,49): number analyzed (Participants) | 46 | 47 | 49
  Week 4 (n=46,47,49) | -0.7 (2.67) | -0.6 (2.62) | -0.6 (2.51)
  Week 8 (n=47,45,45): number analyzed (Participants) | 47 | 45 | 45
  Week 8 (n=47,45,45) | -1.2 (3.51) | -0.8 (2.46) | -0.9 (2.85)
  Week 12 (n=46,45,47): number analyzed (Participants) | 46 | 45 | 47
  Week 12 (n=46,45,47) | -0.9 (3.33) | -0.5 (2.19) | -1.5 (3.14)

13. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week of Tear Production - Schirmer Test (mm) (Oculus Dexter (OD) = Right Eye)
Description: The Schirmer's test was performed without anesthetic. Tear secretion was measured in millimeters based on the length of strip wetted by tears (max score =35 mm/eye). Lower values indicate lower relative amounts of tear secretion (worsening). A negative change from baseline is a positive outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 49 | 47 | 49
mm
  Week 2 (n=49,45,46): number analyzed (Participants) | 49 | 45 | 46
  Week 2 (n=49,45,46) | -1.1 (8.38) | -0.3 (8.62) | -0.3 (7.67)
  Week 4 (n=46,47,49): number analyzed (Participants) | 46 | 47 | 49
  Week 4 (n=46,47,49) | -0.3 (7.45) | -1.4 (7.85) | 0.1 (7.40)
  Week 8 (n=47,43,45): number analyzed (Participants) | 47 | 43 | 45
  Week 8 (n=47,43,45) | 0.0 (8.04) | -1.7 (9.89) | -1.4 (8.45)
  Week 12 (n=46,45,47): number analyzed (Participants) | 46 | 45 | 47
  Week 12 (n=46,45,47) | -0.7 (7.79) | -0.9 (7.02) | 0.9 (7.77)

14. Secondary Outcome: Ocular Surface Parameters: Summary Statistics of Change From Baseline by Week of Tear Production - Schirmer Test (mm) (Oculus Sinister (OS) = Left Eye)
Description: as for outcome 13
Time Frame: Baseline, Weeks 2, 4, 8, 12
Population: Participants in the Full Analysis Set with an available value for the outcome measure at baseline and at each timepoint.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 49 | 47 | 49
mm
  Week 2 (n=49,45,46): number analyzed (Participants) | 49 | 45 | 46
  Week 2 (n=49,45,46) | -0.7 (8.98) | -1.5 (7.81) | 0.6 (4.82)
  Week 4 (n=46,47,49): number analyzed (Participants) | 46 | 47 | 49
  Week 4 (n=46,47,49) | 0.7 (7.52) | -2.1 (7.78) | 1.4 (7.59)
  Week 8 (n=47,43,45): number analyzed (Participants) | 47 | 43 | 45
  Week 8 (n=47,43,45) | 0.2 (8.30) | -1.1 (8.71) | -0.7 (6.92)
  Week 12 (n=46,45,47): number analyzed (Participants) | 46 | 45 | 47
  Week 12 (n=46,45,47) | 0.1 (9.51) | -2.2 (8.60) | 1.1 (7.88)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of 119 days (approximately 4 months).
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 50 | 49 | 51
Participants
  Any adverse events | 21 | 12 | 18
  -Any ocular adverse events | 11 | 10 | 10
  -Any non-ocular adverse events | 13 | 4 | 13
  Any serious adverse events | 0 | 0 | 1
  -Any ocular serious adverse events | 0 | 0 | 0
  -Any non-ocular serious adverse events | 0 | 0 | 1
  Any study drug related adverse events | 5 | 5 | 2
  -Any study drug related ocular adverse events | 5 | 5 | 2
  -Any study drug related non-ocular adverse events | 0 | 1 | 0
  Any adverse events leading to study drug discontinuation | 1 | 1 | 1
  -Any ocular adverse events leading to study drug discontinuation | 0 | 1 | 0
  -Any non-ocular adverse events leading to study drug discontinuation | 1 | 1 | 1
  Any study drug related serious adverse events | 0 | 0 | 0
  -Any study drug related ocular serious adverse events | 0 | 0 | 0
  -Any study drug related non-ocular serious adverse events | 0 | 0 | 0
  Death | 0 | 0 | 0

16. Secondary Outcome: Ocular Treatment Emergent Adverse Events, by Primary System Organ Class (SOC) and Preferred Term (PT)
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
  MedDRA Version 26.0 was used for the reporting of adverse events.
Time Frame: as for outcome 15
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 50 | 49 | 51
Participants
  Number of subjects with at least one event | 11 | 10 | 10
  SOC: Eye disorders | 10 | 8 | 10
  -Eye pain | 3 | 0 | 2
  -Dry eye | 2 | 2 | 0
  -Eye pruritus | 2 | 1 | 0
  -Dry age-related macular degeneration | 1 | 0 | 0
  -Eye discharge | 1 | 2 | 1
  -Eye irritation | 1 | 1 | 1
  -Vision blurred | 1 | 1 | 1
  -Vitreous detachment | 1 | 0 | 0
  -Blepharitis | 0 | 0 | 1
  -Chalazion | 0 | 0 | 2
  -Conjunctival papillae | 0 | 1 | 0
  -Corneal oedema | 0 | 0 | 1
  -Erythema of eyelid | 0 | 3 | 0
  -Lacrimation increased | 0 | 1 | 0
  -Ocular hyperaemia | 0 | 2 | 1
  -Optic nerve cupping | 0 | 0 | 1
  -Swelling of eyelid | 0 | 1 | 0
  SOC: General disorders and administration site conditions | 0 | 4 | 0
  -Instillation site irritation | 0 | 2 | 0
  -Instillation site pruritus | 0 | 1 | 0
  -Therapy responder | 0 | 1 | 0
  SOC: Immune system disorders | 0 | 1 | 0
  -Drug hypersensitivity | 0 | 1 | 0
  SOC: Infections and infestations | 2 | 0 | 0
  -Hordeolum | 2 | 0 | 0
  SOC: Injury, poisoning and procedural complications | 0 | 0 | 1
  -Corneal abrasion | 0 | 0 | 1
  -Foreign body in eye | 0 | 0 | 1

17. Secondary Outcome: Summary of Non-ocular Treatment Emergent Adverse Events
Description: as for outcome 15
Time Frame: as for outcome 15
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | SAF312 15 mg/mL | SAF312 5mg/mL | SAF312 Placebo
Number analyzed (Participants) | 50 | 49 | 51
Participants | 13 | 4 | 13

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum timeframe of 119 days (approximately 4 months).
Groups:
- Total: Total
Arm/Group | SAF312 15 mg/mL | SAF312 5 mg/mL | SAF312 Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/51 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 1/51 | 1/150
Other Adverse Events (participants affected / at risk) | 21/50 | 12/49 | 18/51 | 51/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAF312 15 mg/mL (N=50) | SAF312 5 mg/mL (N=49) | SAF312 Placebo (N=51) | Total (N=150)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAF312 15 mg/mL (N=50) | SAF312 5 mg/mL (N=49) | SAF312 Placebo (N=51) | Total (N=150)
Blepharitis (Eye disorders) | 0 | 0 | 1 | 1
Chalazion (Eye disorders) | 0 | 0 | 2 | 2
Conjunctival papillae (Eye disorders) | 0 | 1 | 0 | 1
Corneal oedema (Eye disorders) | 0 | 0 | 1 | 1
Dry age-related macular degeneration (Eye disorders) | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 2 | 0 | 4
Erythema of eyelid (Eye disorders) | 0 | 3 | 0 | 3
Eye discharge (Eye disorders) | 1 | 2 | 1 | 4
Eye irritation (Eye disorders) | 1 | 1 | 1 | 3
Eye pain (Eye disorders) | 3 | 0 | 2 | 5
Eye pruritus (Eye disorders) | 2 | 1 | 0 | 3
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 2 | 1 | 3
Optic nerve cupping (Eye disorders) | 0 | 0 | 1 | 1
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 1 | 3
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Instillation site irritation (General disorders) | 0 | 2 | 0 | 2
Instillation site pruritus (General disorders) | 0 | 1 | 0 | 1
Medical device site irritation (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Therapy responder (General disorders) | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 1 | 3 | 6
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 2 | 0 | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Buttock injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT04630158/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04630158/SAP_001.pdf